CLINICAL TRIAL: NCT02185092
Title: Probiotic Use in Patients With Prior COPD Exacerbation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lost funding
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4258; RSRCH032089 (Other: OUHSC)
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: COPD; Obstructive Lung Disease
Keywords: exacerbations; COPD; pneumonia; probiotic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Pneumonia | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): 1 pill orally daily
  Interventions: Other: Sugar pill
- Lactobacillus GG (Active Comparator): 1 pill (2 x 10x 9 CFU) daily orally
  Interventions: Dietary Supplement: Lactobacillus GG

INTERVENTIONS:
Dietary Supplement: Lactobacillus GG — probiotic supplement
  Other Names: Culturelle
  Arms: Lactobacillus GG
Other: Sugar pill — placebo
  Arms: Sugar Pill

SUMMARY:
The purpose of the study is to examine the hypothesis test that probiotics will reduce the frequency of exacerbation in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to OUMC or VAMC with a COPD exacerbation and pneumonia with underlying COPD will be eligible and screened.
2. Patients seen in VA Chest Medicine clinic, OU Physicians clinic and Pulmonary fellows clinic at PPOB who have had a COPD exacerbation within the last year.
3. Patients over age 18
4. Patients who have a pulmonary function test (PFT) showing COPD within 1 year of enrollment in the study or if the treating physician plans to obtain PFT as part of the patient's care plan.
5. Patients will be considered to have a diagnosis of COPD if they have a FEV1 of less than 80% of predicted and a FVC/FEV1 ratio of less than 0.70 (as defined by GOLD criteria).

Exclusion Criteria:

1. Patients with less than one year of life expectancy from a concomitant diagnosis
2. Any GI motility disorders or previous bowel resection surgery (short gut syndrome)
3. Any patients with decreased immune function or on medication that may decrease immune function (other than low dose steroid or steroid taper).
4. Patients admitted within the last one year with a diagnosis of pancreatitis
5. Patients unable to give consent will not be included in the study.
6. Patients unable to sign consent
7. Patients already on azithromycin daily for COPD exacerbations
8. Patients under department of corrections custody.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
COPD exacerbations | 1 year
  The primary end point will be the number of COPD exacerbations.

SECONDARY OUTCOMES:
Antibiotic Use | 1 year
  Decreased oral or IV antibiotic use

OTHER OUTCOMES:
Systemic Steroid Use | 1 year
  Decreased systemic steroid use

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Allen, MD, Principal Investigator — OUHSC
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No